CLINICAL TRIAL: NCT01515696
Title: Impact of Oral Application of Gastrografin on the Meconium Evacuation in Very Low Birth Weight Infants- a Phase 4 Study
Brief Title: Impact of Oral Application of Gastrografin on the Meconium Evacuation in Very Low Birth Weight Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nadja Haiden,MD (Other)
Responsible Party: Sponsor-Investigator, Nadja Haiden,MD, Assoc.Prof.MD., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 27112001; 2007-000851-33 (EudraCT Number)
Record Dates: First submitted 2012-01-10; First posted 2012-01-24 (Estimated); Results first posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-06

CONDITIONS: Meconium Ileus; Very Low Birth Weight Infant
Keywords: VLBW infant; Meconium; Enteral nutrition; Meconium passage
MeSH Terms: conditions — Meconium Ileus | interventions — Diatrizoate Meglumine; Diatrizoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gastrografin (Active Comparator): infants receive 3ml/kg Gastrografin + 6ml/kg sterile water
  Interventions: Drug: Gastrografin
- Sterile water (Placebo Comparator): infants receive 9ml/kg sterile water
  Interventions: Drug: Sterile water

INTERVENTIONS:
Drug: Gastrografin — Patients will receive 3ml Gastrografin + 6ml sterile water/kg as a single dose via a nasogastric tube during the first 24 hours of life.
  Other Names: Diatrizoate Meglumine, Diatrizoate Sodium; NDA-011245
  Arms: Gastrografin
Drug: Sterile water — Patients will receive 9ml/kg sterile water as a single dose via a nasogastric tube during the first 24 hours of life.
  Other Names: Sterile water (ANDA) #077393
  Arms: Sterile water

SUMMARY:
Gastrografin is a radiopaque contrast agent for the gastrointestinal tract (GIT) which can be applied orally or rectally. In neonatal intensive care, Gastrografin is used to detect otherwise radiologically invisible perforations or an insufficient GIT anastomosis after surgery. Furthermore it is used for the treatment of meconium ileus. Gastrografin has a strong osmotic effect and leads to water influx into the intestine lumen. Thereby the peristaltic movement is accelerated and the premature infant excretes stool during the hours following application. Therefore Gastrografin might be effective to mobilize meconium from small bowel and deep parts of the colon. The investigators hypothesized that enteral application of Gastrografin accelerates meconium evacuation in premature infants, and thereby enhances feeding tolerance in this population.

DETAILED DESCRIPTION:
In premature infants the establishment of proper gastrointestinal function is challenging and often associated with delayed meconium passage. Meconium evacuation depends on gestational age and birthweight: the more immature an infant is, the later meconium passage starts and the longer meconium passage lasts. The mean duration of meconium evacuation in premature infants with a gestational age below 30 weeks is 8 days, while mature infants excrete their meconium in 2 days. The obstruction of deep intestinal segments by tenacious, sticky meconium frequently leads to gastric residuals, a distended abdomen and delayed food passage. The time lag to full enteral feedings is extended, the probability to acquire infections due to intravenous access for parenteral nutrition increases and the hospital stay of the infant is prolonged. However, the relation between meconium passage and feeding tolerance remains controversial. While one study showed that there is little concordance between first meconium passage and feeding tolerance, an other one showed that rapid and complete excretion of meconium is crucial for oral feeding tolerance and has a positive effect on it. Recently, the investigators performed a prospective randomized trial to determine, whether repeated prophylactic applications of small volume glycerin enemas accelerate passage of meconium in very low birth weight (VLBW) infants. Disappointingly, application of enemas did not accelerate meconium evacuation. A possible reason for the ineffectiveness of glycerin enemas is that the volume used was too small to mobilize tenacious meconium sufficiently from the colon and small bowel.

Gastrografin is a radiopaque contrast agent for the gastrointestinal tract (GIT) which can be applied orally or rectally. In neonatal intensive care, Gastrografin is used to detect otherwise radiologically invisible perforations or an insufficient GIT anastomosis after surgery. Furthermore it is used for the treatment of meconium ileus. Gastrografin has a strong osmotic effect and leads to water influx into the intestine lumen. Thereby the peristaltic movement is accelerated and the premature infant excretes stool during the hours following application. Therefore Gastrografin might be more effective to mobilize meconium from small bowel and deep parts of the colon. The investigators hypothesized, that enteral application of Gastrografin accelerates meconium evacuation in premature infants, and thereby enhances feeding tolerance in this population. The objective of the present study is to determine whether the enteral application of the osmotic contrast agent Gastrografin® accelerates complete meconium excretion and improves feeding tolerance in very low birth weight infants.

ELIGIBILITY:
Inclusion Criteria:

* premature infants with a birthweight < 1500g and a gestational age < 32 weeks

Exclusion Criteria:

* major congenital disorders
* chromosomal aberrations
* systemic metabolic disease and
* pre-existing gastrointestinal abnormalities (i.e. Morbus Hirschsprung)
* pre-existing conditions of severe hypotension

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2007-10; Primary Completion 2010-10 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadja Haiden, MD, Principal Investigator — Medical university of Vienna, Department of Pediatrics

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 year study period 789 infants were eligible for enrollment in the study
Pre-assignment Details: Six hundred ninety-three infants were excluded for the following reasons: informed consent was not obtained in time(n = 660), parental refusal (n = 21), and 12 infants died before randomization.
Groups:
- Gastrografin: infants received 3ml/kg Gastrografin + 6ml/kg sterile water once during the first 24 hours of life via gastric tube
- Sterile Water: infants received 9ml/kg sterile water once during the first 24 hours of life via gastric tube
Period: Overall Study
Arm/Group | Gastrografin | Sterile Water
Started | 47 | 49
Completed | 39 | 39
Not Completed | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gastrografin | Sterile Water | Total
Number analyzed (Participants) | 47 | 49 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 47 | 49 | 96
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 20 | 47
  Male | 20 | 29 | 49
Region of Enrollment [Number; unit: participants]
  Austria | 47 | 49 | 96
birthweight [Median (Full Range); unit: grams] | 870 (0) [490 to 1440] | 900 (0) [480 to 1414] | 879 (0) [480 to 1440]

OUTCOME MEASURES:

1. Primary Outcome: Time to Complete Meconium Evacuation in Days
Description: Time to complete meconium evacuation in days of life until the complete meconium evacuation from birth up to 40 days of life
Time Frame: days of life until until the complete meconium evacuation from birth up to 40 days of life
Population: per protocol
Measure: Median (Full Range); unit: days of life
Arm/Group | Gastrografin | Sterile Water
Number analyzed (Participants) | 39 | 39
days of life | 7 [3 to 16] | 8 [1 to 24]
Statistical Analysis 1: Comparison: Gastrografin vs Sterile Water; Test type: Superiority or Other; p = 0.61, Wilcoxon (Mann-Whitney); Median Difference (Net) = 1

2. Secondary Outcome: Feeding Tolerance- Full Enteral Feedings
Description: full enteral feeding is defined in days of life from birth until an an infant tolerates an enteral feeding volume of 140ml/kg
Time Frame: days of life from birth until an infant tolerates en enteral feeding volume of 140 ml/kg
Population: per protocol
Measure: Median (Full Range); unit: days
Arm/Group | Gastrografin | Sterile Water
Number analyzed (Participants) | 39 | 39
days | 19 [10 to 68] | 26.5 [9 to 109]
Statistical Analysis 1: Comparison: Gastrografin vs Sterile Water; Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 7.5

3. Post Hoc Outcome: Necrotizing Enterocolitis
Description: necrotizing enterocolitis stage 2a after Bell
Time Frame: End of study
Measure: Number; unit: participants
Arm/Group | Gastrografin | Sterile Water
Number analyzed (Participants) | 39 | 39
participants | 8 | 3
Statistical Analysis 1: Comparison: Gastrografin vs Sterile Water; Test type: Superiority or Other; p > 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: from birth until discharge of the infant with a maximum of 5 months
Arm/Group | Gastrografin | Sterile Water
Serious Adverse Events (participants affected / at risk) | 43/47 | 42/49
Other Adverse Events (participants affected / at risk) | 5/47 | 6/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gastrografin (N=47) | Sterile Water (N=49)
intraventricular haemorrhage (Nervous system disorders) | 3 (3) | 3 (3) — intraventricular haemorrhage grade 3 and 4 according the definition of papillae et al
necrotizing enterocolitis (Gastrointestinal disorders) | 10 (10) | 4 (4) — necrotizing enterocolitis stage II or more according to Bell
persistent ductus arteriosus (Cardiac disorders) | 22 (22) | 28 (28)
death (Congenital, familial and genetic disorders) | 8 (8) | 7 (7) — death because of immaturity and associated complications like multiple organ failure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gastrografin (N=47) | Sterile Water (N=49)
culture proven sepsis (Infections and infestations) | 5 (5) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No